CLINICAL TRIAL: NCT04295928
Title: Mise en Place d'un Plan Pharmaceutique Personnalisé Chez Les Patients transplantés rénaux ou hépatiques : Essai randomisé en Cluster de Type Stepped-wedge.
Brief Title: Establishment of a Personalized Pharmaceutical Plan in Renal or Hepatic Transplant Patients
Acronym: GREPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Unité d'Epidémiologie des Données cliniques en Centre-Val de Loire (EpiDcliC) (Unknown); Unité d'Evaluation Médico-Economique (UEME) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: DR190061-GREPH; 2019-A01723-54 (Registry Identifier: ID RCB); 920070 (Registry Identifier: CNIL)
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Personalized Pharmaceutical Plan After Transpantation
Keywords: Therapeutic adherence; Immunosuppressive treatments; Transplantation; Liver; Kidney; Personalized Pharmaceutical Plan; Community-hospital link
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Cluster Stepped-wedge; Inclusions per cluster: Control period->Leeadin period->Interventionnal period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Implementation of a personalized pharmaceutical plan with a view to increasing the patient's therapeutic education in the hospital and in the community (entrance and discharge reconciliation, 3 pharmaceutical interviews in the hospital, strengthening of the community-hospital link , 3 outpatient pharmaceutical consultations)
  Interventions: Behavioral: PPP
- Usual care period (No Intervention): No changes to usual center practices

INTERVENTIONS:
Behavioral: PPP — Personalized Pharmaceutical Plan on therapeutic adherence to immunosuppressive treatments after the transplantation
  Arms: Intervention

SUMMARY:
The main objective of the study is to evaluate the impact of the Personalized Pharmaceutical Plan on the therapeutic adherence to immunosuppressive treatments one year after liver or kidney transplantation.

DETAILED DESCRIPTION:
In 2016, 3,615 renal transplantations (RT) were performed in France. RT is indicated for end-stage renal failure, especially in dialysis patients. The average cost of a year of dialysis is 60,000 €, and that of a kidney transplantation according to the GHS tariff of 20,000 € (excluding preparation of the patient for the transplantation, drugs and post-transplantation follow-up).

In 2016, 1,322 liver transplantations (LT) were performed in France. Indications for LT are mainly acute or chronic hepatic insufficiency and liver tumors. LT is the only therapeutic solution for these patients because there is no such alternative as dialysis in nephrology. According to the DRG (Diagnosis Related Group) tariff, the average cost of a LT is about 35,000€ (excluding preparation for transplantation, drugs and post-transplantation follow-up).

If kidney and liver transplantations allow the patient to return to a life close to normal, with graft survival at one year of 84% for the liver and 91% for the kidney, these is constrained by taking immunosuppressive treatments (IS). In the last few years, progress has been made both in surgery and in immediate post-transplantation management. Therefore, now, the challenges of transplantation lie in the long-term transplant patients management, that is to say in prevention of transplant organ rejection and of anti-rejection drugs side effects (cardiovascular diseases, cancers, infections). This prevention requires optimal adherence of the patients both to the drug treatment and to the hygieno-dietetic rules. The scarcity of grafts in France makes it necessary to maximize graft survival so as to limit the need for a new transplantation.

In the literature, drug adherence of IS is between 45% and 85%. Among the non-adherence factors identified, there is a lack of a therapeutic education program and the delay with respect to the transplantation (with the spacing of the consultations at the hospital).

The investigators hypothesize that the combination of pharmaceutical follow-up during hospitalization, coupled with a strengthened hospital-community link, is central to patient adherence, and therefore to patient and graft survival.

The French Society of Clinical Pharmacy (SFPC) established in 2017 a new model of clinical pharmacy. The latter is based (apart from the regulatory activity of prescriptions analysis), on the implementation of a Personalized Pharmaceutical Plan (PPP) corresponding to a management adapted to the patient's path by proposing best possible medication history, pharmaceutical interviews, dedicated pharmaceutical outpatient consultations and therapeutic education. These actions must be carried out both at the hospital and at the local pharmacy.

Most often, the post-transplantation follow-up is done by the transplant center or for some cases (especially for the liver) by expert centers closer to the patient's home but often quite far from the transplant team. Primary care teams have little or no integration into the care of these patients. This is why the community pharmacist, in collaboration with the transplant team, could be a relay close to the patient ensuring continuity, repetition of messages and follow-up as soon as the post-transplantation consultations spread out.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient having given his free, informed and express consent
* Patient with a kidney or liver transplantation performed in the 10 participating university hospital centers
* Patient speaking french
* Patient whose main residence is in France and has no project of moving during the study period
* Patient declaring to attend the same pharmacy
* Social insured patient

Exclusion Criteria:

* Patient protected: safeguard of justice, curatorship, tutelage
* Patient having a double liver / kidney transplantation with a center not participating in the study
* Patients with a double organ transplantation kidney /hart
* Patient already transplanted regardless of the organ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1716 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adhesion | 1 year after transplantation
  The Investigator will consider that a patient is in therapeutic adhesion thanks to two methods : use of the BAASIS® questionnaire (if answer <1 for at least one of the 4 questions in the score, the patient will be considered as a non-adherent) and use of the health insurance data from the national health data system (checking that 100% of the days are covered by possession of immunosuppressive drugs)

SECONDARY OUTCOMES:
Drug adherence of all chronic treatments prescribed to the patient (except immunosuppression (IS) drug) | 1 year after transplantation
  Drug adherence of all chronic treatments prescribed to the patient (except immunosuppression (IS) drug) measured by the EvalObs® scale (graduation from 0 to 15)
Knowledge of hygienic-dietetic rules and drug intake modalities | 1 year after transplantation
  Knowledge of hygienic-dietetic rules and drug intake modalities assessed using an questionnaire ( scale from 1-9)
Occurrence of adverse effects | At month 1,month 3, and 12 months after transplantation
  Search for the occurrence of adverse events related to IS (diabetes, hypertension, weight gain, tremor, leukopenia, thrombocytopenia,...) during medical and pharmaceutical consultations.
Fate of the graft | 1 year and 3 years after transplantation
  Study of the fate of the graft (rejection, rejection episodes)
Assessing patient, medical, and community pharmacist satisfaction | 1 year after transplantation
  Assessing patient, medical, community pharmacist and trial satisfaction (thanks to a 5-level Likert scale) with the system implemented
Assessment of potential release risk by measuring the coefficient of variation (CV) of anticalcineurin doses | 3 years after transplantation
  A patient with a CV greater than 30% will be considered to be at higher risk of rejection
For kidney transplantation : testing for anti-HLA antibodies | 1 year and 3 years after transplantation
  Anti-HLA antibodies are known to be responsible for rejection in kidney transplants: search for anti-HLA antibodies directed against the donor one and three years after the transplant by Elisa technique
Determining the efficiency of the implementation of the PPP | 1 year after transplantation
  Determining the efficiency of the implementation of this PPP in 3 different ways: by determining the cost per QALY gained at 1 year, the cost per additional patient adherent at 1 year and the cost per first functional graft in additional living patient (living patient, carrying their first graft and functional graft) at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xavier POURRAT, PhD, Study Director — University Hospital of TOURS
Locations (12):
- France (12):
  - CHU-BREST - Pharmacie clinique La Cavale Blanche, Brest
  - APHM - Service de Pharmacie Clinique; Hôpital de la Timone, Marseille
  - APHM Service Pharmacie- Hôpital de la Conception, Marseille
  - CHU-Montpellier Service Pharmacie Lapeyronie, Montpellier
  - CHU-NANTES Service de Pharmacie, Nantes
  - CHU-POITIERS Service de Pharmacie, Poitiers
  - CHU-REIMS Service de Pharmacie -Robert Debré, Reims
  - CHU-RENNES Pôle Pharmacie, Unité de pharmacie clinique, Rennes
  - CHU-STRASBOURG Service Pharmacie, Hôpital Hautepierre, Strasbourg
  - CHU-TOULOUSE Pôle Pharmacie PURPAN, Toulouse
  - CHU-TOURS Hôpital Bretonneau, Tours
  - CHU-TOURS-Hôpital TROUSSEAU, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pourrat X, Berthy E, Dupuis A, Barbier L, Buchler M, Guillon LG, Monmousseau F, Ruspini E, Salame E, Houdard SB, Giraudeau B. Implementing a personalized pharmaceutical plan in kidney or liver transplant patients: study protocol for a stepped-wedge cluster randomized trial (GRePH). Trials. 2021 Nov 8;22(1):782. doi: 10.1186/s13063-021-05749-w. PMID 34749777